CLINICAL TRIAL: NCT05599529
Title: A Retrospective Cohort Study of Differential Attainment, COVID-19 and Chaos: Taking the Difference Out of a Terrible Trinity
Brief Title: A Retrospective Cohort Study of Differential Attainment, COVID-19 and Chaos
Status: Completed | Type: Observational
Sponsor: Health Education and Improvement Wales (Other)
Responsible Party: Sponsor
Other Study IDs: CST_COVID_Outcomes
Record Dates: First submitted 2022-10-25; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Surgery; COVID-19
Keywords: Core Surgical Training; Differential Attainment; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-COVID
  Interventions: Other: Differential attainment
- Peri-COVID
  Interventions: Other: Differential attainment

INTERVENTIONS:
Other: Differential attainment — Differential attainment related to covid, ethnicity and international graduate status

SUMMARY:
A retrospective cohort study of Differential Attainment, COVID and Chaos: taking the difference out of a terrible trinity

DETAILED DESCRIPTION:
Background: This study aimed to evaluate Core Surgical Training (CST) Differential Attainment (DA) related to COVID-19 and gender in three ethnic cohorts: White UK (WUKG), Black & Minority Ethnic UK (BMEUKG), and International Medical Graduates (IMG). The hypothesis was that COVID-19 adversely influenced CST outcome.

Methods: Anonymised 234 CST and 37 IST records (152 WUKG, 81 BMEUKG, 38 IMG) in a UK Statutory Education Body (SEB) were examined. Primary effect measures were: Annual Review of Competency Progression Outcome (ARCPO), MRCS pass, and National Training Number (NTN) appointment.

ELIGIBILITY:
Inclusion Criteria:

* CST

Exclusion Criteria:

* Not completed training

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Core Surgical Trainees in HEIW 2014-2022
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Successful outcome in Membership of the Royal College of Surgeons examination | 2014-2022
Succesful Annual Review of Competence Progression Outcome | 2014-2022
National Training Number Appointment | 2014-2022

SECONDARY OUTCOMES:
Operative Logbook Volume | 2014-2022
Attrition rate | 2014-2022

CONTACTS AND LOCATIONS:
Overall Officials: Osian James, Principal Investigator — HEIW
Locations (1):
- HEIW School of Surgery, Nantgarw, Caerdydd, United Kingdom

REFERENCES:
- [Derived] James OP, Mellor K, Luton O, Robinson DBT, Walsh L, Hemington-Gorse S, Egan RJ, Lewis WG. A retrospective cohort study of differential attainment, COVID and chaos: taking the difference out of a terrible trinity. Int J Surg. 2023 Aug 1;109(8):2359-2364. doi: 10.1097/JS9.0000000000000488. PMID 37222671